CLINICAL TRIAL: NCT04588792
Title: Nebulized Furosemide for Pulmonary Inflammation in Intubated Patients With COVID-19 - A Phase 2/3 Study
Brief Title: Furosemide as Supportive Therapy for COVID-19 Respiratory Failure
Acronym: FaST-1
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of recruitment due to decline in critically ill Covid-19 patients
Sponsor: Dr. John Muscedere (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor-Investigator, Dr. John Muscedere, Professor of Medicine, Queen's University, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FaST-1
Record Dates: First submitted 2020-10-14; First posted 2020-10-19 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Covid19; Respiratory Failure
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaled Furosemide (Experimental): 40 mg furosemide per dose, given by nebulization (4 mL of 10 mg/mL furosemide in 0.9% saline solution) over 30 mins four times daily (Q6H) for up to 28 days
  Interventions: Drug: Nebulized Furosemide
- Nebulized Saline (Placebo Comparator): Placebo, given by nebulization (4 mL of 0.9% saline solution) over 30 mins four times daily (Q.I.D.) for up to 28 days
  Interventions: Drug: Nebulized Saline

INTERVENTIONS:
Drug: Nebulized Furosemide — Furosemide administered by nebulization through the ventilator circuit
  Arms: Inhaled Furosemide
Drug: Nebulized Saline — Saline administered by nebulization through the ventilator circuit
  Arms: Nebulized Saline

SUMMARY:
This double-blind, placebo-controlled, randomized, parallel-group phase 2/3 study will study the utility of nebulized furosemide for pulmonary inflammation in Intubated, mechanically ventilated Patients with COVID-19.

DETAILED DESCRIPTION:
This double-blind, placebo-controlled, randomized, parallel-group phase 2/3 study will study the utility of nebulized furosemide for pulmonary inflammation in Intubated, mechanically ventilated Patients with COVID-19. The primary objective of the study is to establish the efficacy and safety of nebulized furosemide for the treatment of respiratory failure secondary to COVID-19 infection requiring invasive mechanical ventilation. The secondary objective is to delineate the anti-inflammatory properties of furosemide in COVID- 19 patients using pharmacokinetic / pharmacodynamic analysis. The duration of the intervention will be up to 28 days of intervention and patients will be followed till 60 days post randomization. Participants will be randomized to either: Intervention Group: 40 mg furosemide per dose, given by nebulization (4 mL of 10 mg/mL furosemide in 0.9% saline solution) over 30 mins four times daily (Q6H) for up to 28 days OR Control Group: placebo, given by nebulization (4 mL of 0.9% saline solution) over 30 mins four times daily for up to 28 days. One hundred and forty-four (144) evaluable patients will be enrolled in the Phase 2 study. If evidence of efficacy is found in the Phase 2 portion, these patients will be enrolled in the Phase 3 study which aims to recruit 640 patients total (496 additional patients to the phase 2 patients).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with respiratory failure secondary to COVID-19 (SARS-CoV-2) infection/pneumonia requiring invasive mechanical ventilation
2. Duration of mechanical ventilation less than 48 hours as measured from the time of randomization
3. If female, must not be pregnant at the time of enrollment as determined by a serum or urine pregnancy test

Exclusion Criteria:

1. Known history of severe chronic pulmonary disease (e.g., preinfection requirement for home oxygen therapy or presence of chronic hypercapnia (PaCO2< 50 mm Hg); mild -moderate disease is still eligible in the absence of chronic hypercapnia or need for chronic oxygen therapy)
2. In the opinion of the PI, unlikely to survive for >48 hours from time of enrollment
3. Enrollment in another trial of anti-inflammatory therapies for COVID-19.
4. Known allergy to furosemide or sulfonamide agents

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Improvement in pulmonary gas exchange | Study Day 6
  Improvement in oxygenation as determined by a standardized PaO2/FiO2 ratio
Requirement for mechanical ventilation | Baseline to day 28
  Number of ventilator-free days in the first 28 days after enrollment

SECONDARY OUTCOMES:
Mortality | Day 60 post enrollment
  All Cause
Requirement for supplemental oxygen | To day 28 post enrollment
  Number of days of alive and not requiring supplemental oxygen
Duration of ICU Stay | Up to 60 days post enrollment
  Duration of ICU Stay
Length of hospitalization | Up to 60 days post enrollment
  Length of hospitalization
Adverse events | Up to 60 days post enrollment
  Incidence of serious adverse events: incorporated as trial outcomes, defined a priori, in accordance with guidelines for academic ICU drug trials
Inhalation adverse events | Up to day 28
  Adverse events during the nebulization of furosemide

OTHER OUTCOMES:
Serum levels of furosemide | Up to day 28
  Serum levels of furosemide every 7 days until the completion of therapy
Electrolyte abnormalities | Up to day 28
  Altered electrolytes on routine testing (frequency of hypokalemia (< 3.0 meq/L), hypernatremia (> 150 meq/L) or increased bicarbonate levels (>30 meq/L) during the ICU stay
Cytokine levels | Up to day 28
  Levels of serum inflammatory cytokines (IL-6, IL-8, TNF-α) at baseline prior to first dose of intervention, day 7, and the completion of therapy

CONTACTS AND LOCATIONS:
Overall Officials: John Muscedere, MD, Principal Investigator — Queens University
Locations (4):
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - Dalhousie University, Halifax, Nova Scotia
  - Kingston Health Sciences Center, Kingston, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brennecke A, Villar L, Wang Z, Doyle LM, Meek A, Reed M, Barden C, Weaver DF. Is Inhaled Furosemide a Potential Therapeutic for COVID-19? Am J Med Sci. 2020 Sep;360(3):216-221. doi: 10.1016/j.amjms.2020.05.044. Epub 2020 Jun 1. PMID 32622469
- [Background] Wang Z, Wang Y, Vilekar P, Yang SP, Gupta M, Oh MI, Meek A, Doyle L, Villar L, Brennecke A, Liyanage I, Reed M, Barden C, Weaver DF. Small molecule therapeutics for COVID-19: repurposing of inhaled furosemide. PeerJ. 2020 Jul 7;8:e9533. doi: 10.7717/peerj.9533. eCollection 2020. PMID 32704455